CLINICAL TRIAL: NCT00002197
Title: 1592U89 Open-Label Protocol for Pediatric Patients With HIV Infection.
Brief Title: A Study of 1592U89 in HIV-Infected Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 238E; CNAA3007
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-12

CONDITIONS: HIV Infections
Keywords: HIV-1; CD4 Lymphocyte Count; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; abacavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir

INTERVENTIONS:
Drug: Abacavir sulfate

SUMMARY:
The purpose of this study is to see if it is safe to give 1592U89 to children (aged 6 months until 14th birthday) with advanced HIV infection who have few treatment options available. The study also examines the effect 1592U89 has on the levels of HIV in the blood.

DETAILED DESCRIPTION:
This is an open-label, non-randomized study. All patients will be treated with 1592U89. Additionally, since optimal therapy usually includes the combined use of 2 or more antiretroviral agents in advanced patients, other novel antiretroviral therapies may be accessed through commercial means or via compassionate use programs. NOTE: 1592U89 should not be administered as a single new agent added to a failing treatment regimen.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Intravenous immunoglobulin G.
* Erythropoietin, granulocyte colony stimulating factor and granulocyte macrophage colony stimulating factor, for the management of hematologic toxicity.

Patients must have:

* Documented HIV infection.
* High risk for disease progression or mortality as defined by either of the following:
* Viral load > 100,000 copies/ml and CD4 cells < 15% of total lymphocyte count despite at least 4 weeks of therapy with commercially available antiretrovirals or as a result of no therapy due to treatment-limiting toxicity of ZDV, 3TC, and ddI; or HIV-associated encephalopathy refractory to ZDV-containing regimen.
* No access to any 1592U89 pediatric study where the patient could qualify for inclusion.
* Parent or legal guardian with the ability to understand and provide written consent for the patient to participate in the trial. Study patients over 13 years should also give written informed consent whenever possible.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* In the investigator's opinion, the patient is unlikely to comply with the requirements of the study.
* Renal failure requiring dialysis.
* Hepatic failure evident by Grade 3 or 4 hyperbilirubinemia and AST > 10 X upper limits of normal.
* Life-threatening infection or other chronic disease that may interfere with taking 1592U89 or compromise the patient's safety.

Patients with the following prior conditions are excluded:

Documented hypersensitivity to 1592U89 or any other nucleoside analogue.

See Inclusion - General Criteria.

Ages: 6 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States